CLINICAL TRIAL: NCT01712984
Title: Immunogenicity and Safety Trial of Quadrivalent Influenza Vaccine Administered by Intradermal Route in Adult Subjects Aged 18 Through 64 Years
Brief Title: Study of Intradermal Quadrivalent Influenza Vaccine in Adults Aged 18 Through 64 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QID01; U1111-1124-8066 (Other: WHO)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Influenza; Fluzone® Intradermal vaccine; Influenza Virus Vaccine USP Quadrivalent; Influenza Virus Vaccine USP Trivalent Types A and B
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- QIV ID Vaccine Group (Experimental): Participants will receive the intradermal quadrivalent influenza vaccine
  Interventions: Biological: Influenza Virus Vaccine USP Quadrivalent, (Zonal Purified Subvirion) 2012 2013 Formulation
- TIV ID1 Vaccine Group (Active Comparator): Participants will receive the trivalent influenza vaccine containing the B strain from the primary (Yamagata) lineage
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone® Intradermal
- TIV ID2 Group (Active Comparator): Participants will receive the intradermal trivalent influenza vaccine containing B strain from the alternate (Victoria) lineage
  Interventions: Biological: Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone Intradermal

INTERVENTIONS:
Biological: Influenza Virus Vaccine USP Quadrivalent, (Zonal Purified Subvirion) 2012 2013 Formulation — 0.1mL, Intradermal
  Other Names: QIV ID
  Arms: QIV ID Vaccine Group
Biological: Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone® Intradermal — 0.1mL, Intradermal
  Other Names: Fluzone® Intradermal
  Arms: TIV ID1 Vaccine Group
Biological: Influenza Virus Vaccine USP Trivalent Types A and B (Zonal Purified Subvirion) Fluzone Intradermal — 0.1mL, Intradermal
  Other Names: Fluzone® Intradermal
  Arms: TIV ID2 Group

SUMMARY:
The aim of the study is to demonstrate safety and immunogenicity of the quadrivalent influenza intradermal (QIV-ID) vaccine compared to the trivalent influenza vaccine (TIV) containing the B strain from the primary (Yamagata) lineage (TIV-ID1) and the trivalent influenza vaccine containing B strain from the alternate (Victoria) lineage (TIV-ID2) vaccines in producing protection against four strains of influenza virus.

Primary Objective:

* To demonstrate that QIV-ID induces an immune response (as assessed by hemagglutination inhibition (HAI) geometric mean titers (GMTs) and seroconversion rates) that is non-inferior to responses induced by TIV-ID1 and TIV-ID2 for the 4 virus strains at 28 days post-vaccination.

Secondary Objectives:

* To demonstrate that each B strain in QIV-ID induces an immune response (as assessed by HAI GMTs and seroconversion rates) that is superior to the response induced by the TIV-ID that does not contain the corresponding B strain.
* To describe the rate of post-vaccination seroprotection induced by QIV-ID and TIV-ID.
* To describe post-vaccination immunogenicity stratified by age (18-49 years and 50-64 years), race, ethnicity, gender, previous vaccination status, and baseline seropositivity status.
* To describe the safety profile for subjects who receive QIV-ID and TIV-ID.

Observational Objectives:

* To demonstrate non-inferiority of QIV-ID compared to TIV-ID in terms of all Grade 2 or Grade 3 solicited systemic reactions combined
* To demonstrate non-inferiority of QIV-ID compared to TIV-ID in terms of all Grade 3 solicited injection site reactions combined.

DETAILED DESCRIPTION:
All participants will receive a single dose of their assigned vaccine on Day 0. A subset of the participants will be assessed for immunologic response on Day 0 before vaccination and Day 28 after vaccination. All subjects will be monitored for safety for up to 6 months after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 through 64 years on the day of inclusion
* Informed consent form (ICF) has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures. Exclusion Criteria:
* Subject is pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination and until at least 4 weeks after vaccination)
* Participation at the time of trial enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial vaccination
* Vaccination against influenza in the past 6 months
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* History of thrombocytopenia
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion
* Identified as an Investigator or employee of the Investigator or trial center with direct involvement in the proposed trial, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed trial
* Personal or family history of Guillain-Barré Syndrome
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that is stable at the time of vaccination in the absence of therapy, and subjects who have a history of neoplastic disease and who have been disease free for ≥ 5 years.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3360 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (35):
- United States (35):
  - Hoover, Alabama
  - Huntsville, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Chula Vista, California
  - Sacramento, California
  - San Diego, California
  - Milford, Connecticut
  - Coral Gables, Florida
  - Melbourne, Florida
  - Pinellas Park, Florida
  - South Miami, Florida
  - Boise, Idaho
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Kansas City, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Binghamton, New York
  - Rochester, New York
  - Allentown, Pennsylvania
  - Bensalem, Pennsylvania
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Dakota Dunes, South Dakota
  - Austin, Texas
  - Fort Worth, Texas
  - San Angelo, Texas
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Marshfield, Wisconsin

REFERENCES:
- [Background] Gorse GJ, Falsey AR, Ozol-Godfrey A, Landolfi V, Tsang PH. Safety and immunogenicity of a quadrivalent intradermal influenza vaccine in adults. Vaccine. 2015 Feb 25;33(9):1151-9. doi: 10.1016/j.vaccine.2015.01.025. Epub 2015 Jan 19. PMID 25613721
- [Derived] Small RD, Ozol-Godfrey A, Yan L. On the use of nonparametric tests for comparing immunological Reverse Cumulative distribution curves (RCDCs). Vaccine. 2019 Oct 16;37(44):6737-6742. doi: 10.1016/j.vaccine.2019.09.007. Epub 2019 Sep 16. PMID 31537446
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 22 October 2012 to 28 May 2013 at 38 clinic sites in the United States.
Pre-assignment Details: A total of 3360 participants who met all of the inclusion and none of the exclusion criteria were randomized, 3355 received one of the trial vaccines and their data are presented in this report.
Groups:
- QIV ID Vaccine Group: Adults 18 to <65 years of age received a single injection of quadrivalent influenza intradermal (QIV ID) vaccine
- TIV ID1 Vaccine Group: Adults 18 to <65 years of age received a single injection of trivalent influenza vaccine containing the B strain from the primary (Yamagata) lineage (TIV ID1)
- TIV ID2 Vaccine Group: Adults 18 to <65 years of age received a single injection of trivalent influenza vaccine containing the B strain from the alternate (Victoria) lineage (TIV ID2)
Period: Overall Study
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Started | 1672 | 837 | 846
Completed | 1656 | 821 | 836
Not Completed | 16 | 16 | 10
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Lost to Follow-up | 8 | 10 | 1
Not completed — Withdrawal by Subject | 6 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group | Total
Number analyzed (Participants) | 1672 | 837 | 846 | 3355
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1672 | 837 | 846 | 3355
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (13.2) | 41.2 (13.5) | 41.9 (13.3) | 41.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1022 | 505 | 528 | 2055
  Male | 650 | 332 | 318 | 1300
Region of Enrollment [Number; unit: Participants]
  United States | 1672 | 837 | 846 | 3355

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers Against the Influenza Virus Antigens Following Vaccination With Either a Quadrivalent Influenza Vaccine or a Trivalent Influenza Vaccine Administered by Intradermal Route
Description: Antibodies against the influenza vaccine virus antigens were measured using a Hemagglutination-inhibition (HAI) assay.
Time Frame: Day 28 post-vaccination
Population: Geometric mean titers against the influenza virus antigens were assessed in the Per-protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Number analyzed (Participants) | 1041 | 539 | 533
Titers
  A/H1N1 (N=1041, 539, 533) | 589 [546 to 636] | 728 [653 to 811] | 635 [568 to 709]
  A/H3N2 (N=1041, 538, 533) | 368 [342 to 397] | 413 [369 to 462] | 447 [401 to 498]
  B/Texas/6/2011 (B1; N=1041, 539, 533) | 105 [99.1 to 112] | 93.5 [85.9 to 102] | 54.0 [49.3 to 59.2]
  B/Brisbane/60/2008 (B2; N=1041, 538, 533) | 136 [128 to 145] | 66.7 [61.0 to 72.9] | 130 [118 to 143]

2. Primary Outcome: Number of Participants With Seroconversion to Influenza Virus Vaccine Antigens Following Vaccination With Either a Quadrivalent Influenza Vaccine or a Trivalent Influenza Vaccine Administered by Intradermal Route
Description: Antibodies against the influenza vaccine virus antigens were measured using a Hemagglutination-inhibition (HAI) assay. Seroconversion was defined as titer< 10 (1/dil) on Day 0 and post injection titer ≥ 40 (1/dil) on Day 28, or titer ≥10 (1/dil) on Day 0 and a ≥4 fold increase in titer (1/dil) on Day 28).
Time Frame: Day 28 post-vaccination
Population: Seroconversion to the influenza virus antigens were assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Number analyzed (Participants) | 1041 | 539 | 533
Participants
  A/H1N1 (N=1041, 539, 533) | 600 | 333 [0 to 0] | 314 [0 to 0]
  A/H3N2 (N=1040, 538, 533) | 608 | 326 [0 to 0] | 314 [0 to 0]
  B/Texas/6/2011 (B1; N=1041, 539, 533) | 580 | 253 [0 to 0] | 131 [0 to 0]
  B/Brisbane/60/2008 (B2; N=1041, 538, 533) | 525 | 119 [0 to 0] | 235 [0 to 0]

3. Secondary Outcome: Geometric Mean Titers Against the Influenza Virus Antigens Before and Following Vaccination With Either a Quadrivalent Influenza Vaccine or a Trivalent Influenza Vaccine Administered by Intradermal Route
Description: Antibodies against the influenza vaccine virus antigens were measured using a Hemagglutination-inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Geometric mean titers against the influenza virus antigens were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Number analyzed (Participants) | 1041 | 539 | 533
Titers
  A/H1N1 Day 0 (N=1041, 539, 533) | 66.3 [59.5 to 73.8] | 65.2 [56.0 to 76.0] | 66.2 [56.9 to 77.0]
  A/H1N1 Day 28 (N=1041, 539, 533) | 589 [546 to 636] | 728 [653 to 811] | 635 [568 to 709]
  A/H3N2 Day 0 (N=1040, 539, 533) | 52.3 [47.5 to 57.5] | 56.5 [49.2 to 64.9] | 55.7 [48.4 to 64.0]
  A/H3N2 Day 28 (N=1041, 538, 533) | 368 [342 to 397] | 413 [369 to 462] | 447 [401 to 498]
  B1 Day 0 (N=1041, 539, 533) | 21.7 [20.5 to 23.1] | 24.7 [22.7 to 27.0] | 22.2 [20.4 to 24.2]
  B1 Day 28 (N=1041, 539, 533) | 105 [99.1 to 112] | 93.5 [85.9 to 102] | 54.0 [49.3 to 59.2]
  B2 Day 0 (N=1041, 539, 533) | 26.8 [25.0 to 28.8] | 29.7 [26.9 to 32.8] | 25.4 [23.0 to 28.1]
  B2 Day 28 (N=1041, 538, 533) | 136 [128 to 145] | 66.7 [61.0 to 72.9] | 130 [118 to 143]

4. Secondary Outcome: Number of Participants With Seroprotection Against Influenza Vaccine Antigens Before (Baseline) and Following Vaccination With Either a Quadrivalent Influenza Vaccine or a Trivalent Influenza Vaccine Administered by Intradermal Route
Description: Antibodies against the influenza vaccine virus antigens were measured using a Hemagglutination-inhibition (HAI) assay. Seroprotection was defined as titer ≥ 40 [1/dil] at baseline and 28 days after vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Seroprotection against influenza virus antigens was assessed in the Per Protocol Analysis Set.
Measure: Number; unit: Participants
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Number analyzed (Participants) | 1041 | 539 | 533
Participants
  A/H1N1 Day 0 (N=1041, 539, 533) | 672 | 334 [0 to 0] | 353 [0 to 0]
  A/H1N1 Day 28 (N=1041, 539, 533) | 1014 | 537 [0 to 0] | 524 [0 to 0]
  A/H3N2 Day 0 (N=1040, 539, 533) | 655 | 340 [0 to 0] | 332 [0 to 0]
  A/H3N2 Day 28 (N=1041, 538, 533) | 1008 | 526 [0 to 0] | 519 [0 to 0]
  B1 Day 0 (N=1041, 539, 533) | 335 | 210 [0 to 0] | 172 [0 to 0]
  B1 Day 28 (N=1041, 539, 533) | 923 | 464 [0 to 0] | 351 [0 to 0]
  B2 Day 0 (N=1041, 539, 533) | 467 | 262 [0 to 0] | 224 [0 to 0]
  B2 Day 28 (N=1041, 538, 533) | 976 | 403 [0 to 0] | 477 [0 to 0]

5. Secondary Outcome: Number of Participants Reporting Solicited Injection Site and Systemic Reactions Following Vaccination With Either a Quadrivalent Influenza Vaccine or a Trivalent Influenza Vaccine Administered by Intradermal Route
Description: Solicited injection site: Pain, Erythema, Swelling, Induration, Ecchymosis, and Pruritus; Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Shivering. Grade 3 injection site: Pain and Pruritus Significant, prevents daily activity; Erythema, Swelling, Induration, and Ecchymosis >100 mm. Grade 3 systemic reactions: Fever ≥39˚C; Headache, Malaise, Myalgia, and Shivering Significant preventing daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site reactions and systemic reactions were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Number analyzed (Participants) | 1672 | 837 | 846
Participants
  Injection site Pain (N=1656,820,838) | 883 | 395 [0 to 0] | 420 [0 to 0]
  Grade 3 Injection site Pain (N=1656,820,838) | 24 | 10 [0 to 0] | 12 [0 to 0]
  Injection site Erythema (N=1656,820,838) | 607 | 279 [0 to 0] | 269 [0 to 0]
  Grade 3 Injection site Erythema (N=1656,820,838) | 7 | 1 [0 to 0] | 3 [0 to 0]
  Injection site Swelling (N=1655,820,838) | 322 | 121 [0 to 0] | 123 [0 to 0]
  Grade 3 Injection site Swelling (N=1655,820,838) | 2 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Induration (N=1656,820,837) | 282 | 111 [0 to 0] | 94 [0 to 0]
  Grade 3 Injection site Induration (N=1656,820,837) | 1 | 0 [0 to 0] | 0 [0 to 0]
  Injection site Ecchymosis (N=1656,820,838) | 43 | 15 [0 to 0] | 15 [0 to 0]
  Grade 3 Injection site Ecchymosis (N=1656,820,838) | 0 | 0 [0 to 0] | 0 [0 to 0]
  Fever (N=1649,819,836) | 13 | 6 [0 to 0] | 4 [0 to 0]
  Grade 3 Fever (N=1649,819,836) | 3 | 1 [0 to 0] | 0 [0 to 0]
  Headache (N=1656,820,838) | 548 | 257 [0 to 0] | 278 [0 to 0]
  Grade 3 Headache (N=1656,820,838) | 53 | 20 [0 to 0] | 15 [0 to 0]
  Malaise (N=1656,820,838) | 459 | 216 [0 to 0] | 255 [0 to 0]
  Grade 3 Malaise (N=1656,820,838) | 49 | 15 [0 to 0] | 21 [0 to 0]
  Myalgia (N=1656,820,838) | 564 | 238 [0 to 0] | 261 [0 to 0]
  Grade 3 Myalgia (N=1656,820,838) | 43 | 12 [0 to 0] | 21 [0 to 0]
  Shivering (N=1656,820,838) | 200 | 85 [0 to 0] | 94 [0 to 0]
  Grade 3 Shivering (N=1656,820,838) | 24 | 5 [0 to 0] | 13 [0 to 0]
  Injection site Pruritus (N=1656,820,838) | 862 | 372 [0 to 0] | 374 [0 to 0]
  Grade 3 Injection site Pruritus (N=1656,820,838) | 47 | 15 [0 to 0] | 19 [0 to 0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 6 months post-vaccination.
Arm/Group | QIV ID Vaccine Group | TIV ID1 Vaccine Group | TIV ID2 Vaccine Group
Serious Adverse Events (participants affected / at risk) | 20/1672 | 14/837 | 11/846
Other Adverse Events (participants affected / at risk) | 883/1672 | 395/837 | 420/846
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QIV ID Vaccine Group (N=1672) | TIV ID1 Vaccine Group (N=837) | TIV ID2 Vaccine Group (N=846)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Dysplasia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | QIV ID Vaccine Group (N=1672) | TIV ID1 Vaccine Group (N=837) | TIV ID2 Vaccine Group (N=846)
Injection site Pain (General disorders) | 883/1656 (883) | 395/820 (395) | 420/838 (420)
Injection site Erythema (General disorders) | 607/1656 (607) | 279/820 (279) | 269/838 (269)
Injection site Swelling (General disorders) | 322/1655 (322) | 121/820 (121) | 123/838 (123)
Injection site Induration (General disorders) | 282/1656 (282) | 111/820 (111) | 94/837 (94)
Injection site Pruritus (General disorders) | 862/1656 (862) | 372/820 (372) | 374/838 (374)
Headache (Nervous system disorders) | 548/1656 (548) | 257/820 (257) | 278/838 (278)
Malaise (General disorders) | 459/1656 (459) | 216/820 (216) | 255/838 (255)
Myalgia (Musculoskeletal and connective tissue disorders) | 564/1656 (564) | 238/820 (238) | 261/838 (261)
Shivering (General disorders) | 200/1656 (200) | 85/820 (85) | 94/838 (94)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.